CLINICAL TRIAL: NCT00000940
Title: A Phase II Trial to Evaluate the Safety and Efficacy of Induction Treatment With Lamivudine Plus Stavudine Plus Abacavir Plus Amprenavir/Ritonavir Followed by Supervised Treatment Interruption in Subjects With Acute HIV Infection or Recent Seroconversion
Brief Title: Five-Drug Anti-HIV Treatment Followed by Treatment Interruption in Patients Who Have Recently Been Infected With HIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACTG 371; 10099 (Registry Identifier: DAIDS ES); ACTG 710 (substudy); ACTG 711 (substudy); ACTG 729 (substudy); ACTG 709 (substudy); AACTG 371
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Stavudine; Amprenavir/Ritonavir; Protease Inhibitors; Lamivudine; VX 478; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; Abacavir Sulfate; Acute Infection; Treatment Interruption
MeSH Terms: conditions — HIV Infections | interventions — Ritonavir; abacavir; amprenavir; Lamivudine; Stavudine

INTERVENTIONS:
Drug: Ritonavir
Drug: Abacavir sulfate
Drug: Amprenavir
Drug: Lamivudine
Drug: Stavudine

SUMMARY:
This study will determine what effect taking a combination of five anti-HIV drugs during the early stage of HIV infection, then temporarily stopping them once or twice, may have on the amount of HIV virus in the blood (viral load). The study will also evaluate the safety and effectiveness of this anti-HIV drug combination.

DETAILED DESCRIPTION:
Acute, primary HIV infection represents a potentially unique opportunity to eradicate the infection. Although plasma viral load rises rapidly, the dominant infecting virus is relatively uniform genetically, and infection may not be fully established in all tissue sites until some time after exposure. Current antiretroviral therapy is able to reduce plasma viral load to unmeasurable levels in established infection. However, there are many questions that remain about the treatment of primary HIV infection. While it is assumed that aggressive antiretroviral regimens are required, it is not known how long they must be continued. It is hoped that after an interval of aggressive therapy, the number of agents could be safely reduced. This study evaluates if viral suppression can be sustained after study therapy is withdrawn.

Participants in this study will receive lamivudine (3TC), stavudine (d4T), abacavir (ABC), amprenavir (APV), and ritonavir (RTV) for at least 52 weeks. During this induction phase, participants will be followed through regular study visits every 4 or 8 weeks. If the participant's viral load and CD4 counts are within study parameters at the end of 52 weeks, the participant will discontinue all antiretroviral medications simultaneously. Participants in the treatment interruption phase will be followed weekly initially, every 2 weeks for 8 weeks, and then every 4 or 8 weeks. Treatment may be restarted if necessary during this phase based on viral load and CD4 counts. If treatment is restarted, the participant will receive 3TC, d4T, APV, and RTV but not ABC. During this reinduction phase, participants will be followed every 4 or 8 weeks.

Depending on viral load and CD4 counts, participants may be eligible for a second treatment interruption phase following the reinduction phase. Participants will once again stop all antiretroviral medications simultaneously and will have the same monitoring as in the first treatment interruption phase. Following this second treatment interruption, participants will be restarted on 3TC, d4T, APV, and RTV and will be evaluated at Weeks 4, 8, 16, and 24, at which time participants go off study.

The length of study participation for individual participants will vary. The length of each phase will be highly dependent on the participant's laboratory parameters. In general, participants will be enrolled in the study for 3 to 4 years. Participants may also enroll in immunology, compartment, pharmacology, and medication compliance substudies.

ELIGIBILITY:
Inclusion Criteria:

* Acute HIV infection (recently infected with HIV or recent seroconversion)
* Karnofsky status of 80 or greater within 14 days prior to study entry
* Acceptable methods of contraception
* Able and willing to give written informed consent

Exclusion Criteria:

* Previously received anti-HIV drugs
* Hepatitis within 30 days prior to study entry
* Pancreatitis within 120 days prior to study entry
* Radiation or chemotherapy within 30 days prior to study entry
* Certain medications within 14 days prior to study entry
* Experimental or investigational therapy within 30 days prior to study entry
* Illness (non-HIV infection, cancer, etc.) at the time of study entry
* Pregnant or breastfeeding

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 1999-05; Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Volberding, MD, Study Chair — San Francisco Veterans Medical Center; Elizabeth Connick, MD, Study Chair — Infectious Disease Division, University of Colorado Health Sciences Center
Locations (18):
- United States (18):
  - USC CRS, Los Angeles, California
  - UCLA CARE Center CRS, Los Angeles, California
  - Ucsd, Avrc Crs, San Diego, California
  - Ucsf Aids Crs, San Francisco, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - SSTAR, Family Healthcare Ctr., Fall River, Massachusetts
  - Washington U CRS, St Louis, Missouri
  - Beth Israel Med. Ctr. ACTU, New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Columbia P&S CRS, New York, New York
  - AIDS Care CRS, Rochester, New York
  - McCree McCuller Wellness Ctr. at the Connection, Infectious Disease Unit, Rochester, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - The Miriam Hosp. ACTG CRS, Providence, Rhode Island

REFERENCES:
- [Background] Ait-Khaled M, Rakik A, Griffin P, Cutrell A, Fischl MA, Clumeck N, Greenberg SB, Rubio R, Peters BS, Pulido F, Gould J, Pearce G, Spreen W, Tisdale M, Lafon S; CNA3003 International Study Team. Mutations in HIV-1 reverse transcriptase during therapy with abacavir, lamivudine and zidovudine in HIV-1-infected adults with no prior antiretroviral therapy. Antivir Ther. 2002 Mar;7(1):43-51. PMID 12008787
- [Background] Garcia F, Plana M, Mestre G, Arnedo M, Gil C, Miro JM, Cruceta A, Pumarola T, Gallart T, Gatell JM. Immunological and virological factors at baseline may predict response to structured therapy interruption in early stage chronic HIV-1 infection. AIDS. 2002 Sep 6;16(13):1761-5. doi: 10.1097/00002030-200209060-00008. PMID 12218387
- [Background] Garcia F, Plana M, Ortiz GM, Bonhoeffer S, Soriano A, Vidal C, Cruceta A, Arnedo M, Gil C, Pantaleo G, Pumarola T, Gallart T, Nixon DF, Miro JM, Gatell JM. The virological and immunological consequences of structured treatment interruptions in chronic HIV-1 infection. AIDS. 2001 Jun 15;15(9):F29-40. doi: 10.1097/00002030-200106150-00002. PMID 11416735
- [Background] Mira JA, Macias J, Nogales C, Fernandez-Rivera J, Garcia-Garcia JA, Ramos A, Pineda JA. Transient rebounds of low-level viraemia among HIV-infected patients under HAART are not associated with virological or immunological failure. Antivir Ther. 2002 Dec;7(4):251-6. doi: 10.1177/135965350200700404. PMID 12553479
- [Background] Tilling R, Kinloch S, Goh LE, Cooper D, Perrin L, Lampe F, Zaunders J, Hoen B, Tsoukas C, Andersson J, Janossy G; Quest Study Group. Parallel decline of CD8+/CD38++ T cells and viraemia in response to quadruple highly active antiretroviral therapy in primary HIV infection. AIDS. 2002 Mar 8;16(4):589-96. doi: 10.1097/00002030-200203080-00010. PMID 11873002
- [Result] Volberding P, Demeter L, Bosch RJ, Aga E, Pettinelli C, Hirsch M, Vogler M, Martinez A, Little S, Connick E; ACTG 371 Team. Antiretroviral therapy in acute and recent HIV infection: a prospective multicenter stratified trial of intentionally interrupted treatment. AIDS. 2009 Sep 24;23(15):1987-95. doi: 10.1097/QAD.0b013e32832eb285. PMID 19696651
- [Result] Connick E, Bosch RJ, Aga E, Schlichtemeier R, Demeter LM, Volberding P; ACTG 709 Team. Augmented HIV-specific interferon-gamma responses, but impaired lymphoproliferation during interruption of antiretroviral treatment initiated in primary HIV infection. J Acquir Immune Defic Syndr. 2011 Sep 1;58(1):1-8. doi: 10.1097/QAI.0b013e318224d0c7. PMID 21637110